CLINICAL TRIAL: NCT00695513
Title: A Phase 1/2 Study on the Effects of BENEO synergy1 on the Generation Rate and Serum Concentration of P-cresol and Related Protein-fermentation Endproducts in Haemodialysis Patients
Brief Title: Inulin and Protein Fermentation in Hemodialysis Patients
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Principal Investigator, Björn Meijers, Dr., Universitaire Ziekenhuizen KU Leuven
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ML3534
Record Dates: First submitted 2008-06-10; First posted 2008-06-12 (Estimated); Last update posted 2011-09-15 (Estimated); Status verified 2011-09

CONDITIONS: Chronic Kidney Disease
Keywords: Food supplement; Haemodialysis
MeSH Terms: conditions — Renal Insufficiency, Chronic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- I (Experimental): BENEO synergy1
  Interventions: Dietary Supplement: BENEO synergy1

INTERVENTIONS:
Dietary Supplement: BENEO synergy1 — 50/50 v/v inulin/oligofructose 10 gram BID
  Other Names: BENEO; Synergy1

SUMMARY:
An important group of protein-bound uremic retention solutes originate from protein fermentation in the colon. P-cresol is a putrefaction metabolite of tyrosine. Indole is generated by fermentation of tryptophan. After absorption, the majority of p-cresol and indole are further metabolised and conjugated to form p-cresylsulphate and indoxyl sulphate. There is clear evidence, both in vitro and in vivo, that accumulation of these conjugated fermentation metabolites in kidney disease is correlated with clinical (cardiovascular) endpoints.

Bacterial protein fermentation can be influenced by altering the colonic microenvironment, influencing the ratio of available carbohydrates to nitrogen, by shortening the colonic transit time or a combination of these. From a theoretical point of view, functional foods, i.e. pro-, pre- and synbiotics, fulfil these criteria.

Prebiotics have been defined as non-digestible food ingredients that beneficially affect the host by selectively stimulating growth, and/or activity, of one or a restricted number of bacteria in the colon. Dietary fibre may suppress the generation of bacterial protein fermentation either by altering the colonic microenvironment or by shortening the colonic transit time. Animal and clinical studies evaluating the effect of dietary fibre supplements on the generation of bacterial fermentation metabolites have provided conflicting results. These discrepancies may be related to specific properties of the dietary fibre investigated. Dietary fibre may impair protein assimilation and the fermentability may vary to a substantial extent.

Inulin and oligofructose have attracted much attention recently as nonabsorbable carbohydrates with prebiotic properties. When inulin and oligofructose were added to a controlled diet, significant increases were noted in colonic bifidobacterial populations, and it has been proposed that these changes promote both colonic and systemic health through modification of the intestinal microflora. Inulin and oligofructose are rapidly and completely fermented by the colonic microflora with the production of acetate and other short-chain fatty acids. In healthy individuals, supplementation with a mixture of inulin and oligofructose was shown to lower p-cresol generation. Although data in healthy volunteers are promising, no data are available in hemodialysis patients.

ELIGIBILITY:
Inclusion Criteria:

* Chronic hemodialysis patients on maintenance dialysis treatment.
* 18 years of age or older
* Written informed consent

Exclusion Criteria:

* Use of pre-/pro-/syn- or antibiotics in preceding 4 weeks.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Estimated)
Dates: Start 2006-03; Primary Completion 2008-07 (Actual); Study Completion 2008-07 (Actual)

PRIMARY OUTCOMES:
Decrease p-cresol serum concentration | 4 weeks

SECONDARY OUTCOMES:
Decreased generation rate of p-cresol | 4 weeks
Decreased serum concentration of related uremic retention solutes | 4 weeks
Change in bowel habits as measured by validated constipation scores | 4 weeks
inflammation (c-reactive protein) | 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Pieter Evenepoel, MD, PhD, Principal Investigator — Universitaire Ziekenhuizen KU Leuven; Bjorn Meijers, MD, Principal Investigator — Universitaire Ziekenhuizen KU Leuven
Locations (1):
- Universitaire Ziekenhuizen Leuven, Leuven, Vlaams-Brabant, Belgium

REFERENCES:
- [Background] Meijers BK, Bammens B, De Moor B, Verbeke K, Vanrenterghem Y, Evenepoel P. Free p-cresol is associated with cardiovascular disease in hemodialysis patients. Kidney Int. 2008 May;73(10):1174-80. doi: 10.1038/ki.2008.31. Epub 2008 Feb 27. PMID 18305466
- [Background] De Preter V, Vanhoutte T, Huys G, Swings J, De Vuyst L, Rutgeerts P, Verbeke K. Effects of Lactobacillus casei Shirota, Bifidobacterium breve, and oligofructose-enriched inulin on colonic nitrogen-protein metabolism in healthy humans. Am J Physiol Gastrointest Liver Physiol. 2007 Jan;292(1):G358-68. doi: 10.1152/ajpgi.00052.2006. Epub 2006 Sep 21. PMID 16990449
- [Derived] Meijers BK, De Preter V, Verbeke K, Vanrenterghem Y, Evenepoel P. p-Cresyl sulfate serum concentrations in haemodialysis patients are reduced by the prebiotic oligofructose-enriched inulin. Nephrol Dial Transplant. 2010 Jan;25(1):219-24. doi: 10.1093/ndt/gfp414. Epub 2009 Aug 19. PMID 19692415